CLINICAL TRIAL: NCT00099502
Title: International, Randomized, Multicenter, Phase IIIb Study in Patients With Relapsing-Remitting Multiple Sclerosis Comparing Over a Treatment Period of at Least 104 Weeks: 1. Double-Blinded Safety, Tolerability, and Efficacy of Betaseron/ Betaferon 250 µg (8 MIU) and Betaseron/-Betaferon 500 µg (16 MIU), Both Given Subcutaneously Every Other Day, and 2. Rater-Blinded Safety, Tolerability, and Efficacy of Betaseron/-Betaferon s.c. Every Other Day With Copaxone 20 mg s.c. Once Daily.
Brief Title: BEYOND: Betaferon/Betaseron Efficacy Yielding Outcomes of a New Dose in Multiple Sclerosis (MS) Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer HealthCare Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91162; EudraCT: 2005-002235-27; 306440; Beyond; NCT00185432 (obsolete NCT alias)
Record Dates: First submitted 2004-12-15; First posted 2004-12-16 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing multiple sclerosis; interferon beta 1b; Betaferon; Betaseron
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b; Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046)
- Arm 2 (Experimental)
  Interventions: Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046)
- Arm 3 (Active Comparator)
  Interventions: Drug: Copaxone

INTERVENTIONS:
Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046) — 250mcg administered s.c. every other day
  Arms: Arm 1
Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046) — 500mcg administered s.c. every other day
  Arms: Arm 2
Drug: Copaxone — 20 mg administered s.c. once daily.
  Arms: Arm 3

SUMMARY:
The purpose of this study is to determine

* whether treatment with Betaferon / Betaseron (interferon beta-1b) 500 micrograms safe, tolerable and more efficacious than treatment with interferon beta-1b 250 micrograms
* whether treatment with Betaferon / Betaseron (interferon beta-1b) tolerable and more efficacious than treatment with Copaxone (Glatiramer Acetate) 20 mg

DETAILED DESCRIPTION:
This study has previously been posted by Berlex, Inc. and Schering AG, Germany. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc., Schering AG Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer HealthCare Pharmaceuticals, Inc.and Bayer Schering Pharma AG, Germany are the sponsors of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients
* Aged 18-55 years
* Diagnosis of RRMS (Relapsing-Remitting Multiple Sclerosis), EDSS score of 0 to 5.0
* Treatment-naive to IFNB or Copaxone

Exclusion Criteria:

* Neurological progression at disease onset or between relapses
* Serious or acute heart diseases
* History of severe depression or suicide attempt
* Serious or acute liver, renal or bone marrow dysfunction
* Monoclonal gammopathy
* Known allergy to Gadolinium-DTPA, to IFNs (Interferons), to glatiramer acetate, to human albumin or to mannitol
* Pregnancy or lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2244 (Actual)
Dates: Start 2003-11; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Hazard ratio for relapses | During the first and during the second 52 weeks

SECONDARY OUTCOMES:
Time to confirmed Expanded Disability Status Score (EDSS) progression | After 52 and after 104 weeks
Magnetic Resonance Imaging (MRI): Change from screening in volume of hypointense lesion on enhanced T1 weighted images | After 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (180):
- United States (55):
  - Birmingham, Alabama
  - Cullman, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Berkeley, California
  - La Jolla, California
  - Sacramento, California
  - San Francisco, California
  - Englewood, Colorado
  - Fort Collins, Colorado
  - Wilmington, Delaware
  - Washington D.C., District of Columbia
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Detroit, Michigan
  - Duluth, Minnesota
  - St Louis, Missouri
  - Henderson, Nevada
  - Reno, Nevada
  - Lebanon, New Hampshire
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Mineola, New York
  - Rochester, New York
  - Stony Brook, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - High Point, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Tualatin, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Seattle, Washington
  - Tacoma, Washington
  - Marshfield, Wisconsin
  - Milwaukee, Wisconsin
- Argentina (4):
  - Buenos Aires, Buenos Aires
  - Buenos Aires, Buenos Aires F.D.
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
- Australia (6):
  - Gosford, New South Wales
  - Kogarah, New South Wales
  - Liverpool, New South Wales
  - Melbourne, Victoria
  - Parkville, Victoria
  - Nedlands, Western Australia
- Austria (4):
  - Sankt Pölten, Lower Austria
  - Graz, Styria
  - Innsbruck, Tyrol
  - Linz
- Belgium (3):
  - Bruxelles - Brussel
  - Leuven
  - Melsbroek
- Brazil (7):
  - Curitiba, Paraná
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - Sao Pulo, São Paulo
  - São Paulo, São Paulo
- Canada (12):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Nepean, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Hull, Quebec
  - Montreal, Quebec
- Aarhus C, Denmark
- Finland (2):
  - Oulu
  - Tampere
- France (12):
  - Rennes, Brittany Region
  - Bordeaux, Gironde
  - Caen
  - Clermont-Ferrand
  - Dijon
  - Lille
  - Lyon
  - Nancy
  - Nantes
  - Nice
  - Nîmes
  - Toulouse
- Germany (19):
  - Heidelberg, Baden-Wurttemberg
  - Bayreuth, Bavaria
  - Regensburg, Bavaria
  - Hennigsdorf, Brandenburg
  - Hamburg, Hamburg
  - Giessen, Hesse
  - Marburg, Hesse
  - Offenbach, Hesse
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Asbach, Rhineland-Palatinate
  - Dresden, Saxony
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Berlin, State of Berlin
- Greece (3):
  - Athens, Attica
  - Thessaloniki, Thessaloniki
  - Athens
- Hungary (5):
  - Budapest
  - Győr
  - Miskolc
  - Pécs
  - Zalaegerszeg
- Ireland (3):
  - Dublin, Dublin 24
  - Cork
  - Dublin
- Israel (7):
  - Ashkelon
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
  - Tel Litwinsky
  - Ẕerifin
- Italy (6):
  - Bari, BA
  - Florence, FI
  - Milan, MI
  - Padua, PD
  - Roma, RO
  - Orbassano, TO
- Riga, Latvia
- Netherlands (3):
  - Nijmegen, Gelderland
  - Breda
  - Sittard
- Bergen, Norway
- Poland (6):
  - Gdansk
  - Katowice
  - Lodz
  - Poznan
  - Warsaw
  - Wroclaw
- Russia (6):
  - Moscow
  - Moskva
  - Nizhny Novogorod
  - Novosibirsk
  - Saint Petersburg
  - Yaroslavl
- Slovenia (2):
  - Ljubljana
  - Maribor
- Spain (3):
  - L'Hospitalet de Llobregat, Barcelona
  - Málaga, Málaga
  - Seville, Sevilla
- Sweden (3):
  - Helsingborg
  - Stockholm
  - Uppsala
- Switzerland (2):
  - Bern, Canton of Bern
  - Sankt Gallen, Canton of St. Gallen
- Ukraine (4):
  - Donetsk
  - Kharkiv
  - Kiev
  - Lviv

REFERENCES:
- [Derived] O'Connor P, Filippi M, Arnason B, Comi G, Cook S, Goodin D, Hartung HP, Jeffery D, Kappos L, Boateng F, Filippov V, Groth M, Knappertz V, Kraus C, Sandbrink R, Pohl C, Bogumil T; BEYOND Study Group; O'Connor P, Filippi M, Arnason B, Cook S, Goodin D, Hartung HP, Kappos L, Jeffery D, Comi G. 250 microg or 500 microg interferon beta-1b versus 20 mg glatiramer acetate in relapsing-remitting multiple sclerosis: a prospective, randomised, multicentre study. Lancet Neurol. 2009 Oct;8(10):889-97. doi: 10.1016/S1474-4422(09)70226-1. Epub 2009 Sep 2. PMID 19729344